CLINICAL TRIAL: NCT06432010
Title: Effect of a Health Check-up Followed by a Collective Coaching on the Quality of Life and Behavioral Change of Retired Persons. A Prospective Study Conducted in Ambulatory.
Brief Title: Quality of Life and Behavioral Change of Retired Persons
Acronym: R-FORM'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Principal investigator, Institut Pasteur de Lille
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-A00408-33
Record Dates: First submitted 2021-10-11; First posted 2024-05-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
Keywords: Nutrition and Physical Activity coaching; Cognition coaching; Longevity; Prevention; Quality of life

STUDY DESIGN:
Intervention Model Description: Exploratory prospective, monocentric, ambulatory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group nutrition and physical activity coaching (Other): Initial health check-up → 7 weeks nutrition and physical activity coaching → 2 telephone follow-ups at 3 and 6 months after → Final health check-up (12 months after)
  Interventions: Other: Group nutrition and physical activity coaching
- Group cognition coaching (Other): Initial health check-up → 7 weeks cognition coaching → 2 telephone follow-ups at 3 and 6 months after → Final health check-up (12 months after)
  Interventions: Other: Group cognition coaching
- control group (No Intervention): The study is controlled by the presence of a control group (non-coaching group). 25 people will be included in the control group. They will only benefit from the initial and final health check-up.

INTERVENTIONS:
Other: Group nutrition and physical activity coaching — Group nutrition and physical activity coaching consists of an initial health check-up, followed by nutrition and physical activity coaching sessions over 7 weeks, 2 telephone follow-ups at 3 and 6 months and finally a final health check-up, 12 months after the end of the group nutrition and physical activity coaching sessions.
  Arms: Group nutrition and physical activity coaching
Other: Group cognition coaching — Group cognition coaching consists of an initial health check-up, followed by cognition coaching sessions over 7 weeks, 2 telephone follow-ups at 3 and 6 months and finally a final health check-up, 12 months after the end of the cognition coaching sessions.
  Arms: Group cognition coaching

SUMMARY:
Researchers have found that the first phase of aging, called "frailty", is insidious, silent and slowly progressive. It begins well before the first signs of aging and possibly before retirement age with physiological reserves that are gradually depleted. Frailty is multifactorial. It is situated between the "robust-vigorous" and "poly-pathological-dependent" stages of aging. This state remains dynamic and above all reversible through screening and awareness of the individual's health determinants as well as motivation to change.

The Longevity Pathway was designed to meet several concrete objectives ranging from improving prevention to advancing research on the topic of longevity and aging well.

This study aims to evaluate the effect of this personalized support on the quality of life of the consultants, but also on many health parameters, 12 months after the end of the proposed coaching.

DETAILED DESCRIPTION:
The study will be carried out on healthy volunteers, retired.

The main objective of the study is to evaluate the effect of a health check-up followed by a collective "coaching" type of support on the quality of life of retired people 12 months after the end of the coaching sessions.

ELIGIBILITY:
Inclusion Criteria:

* Man or Woman;
* Retired;
* Having the desire to change his/her lifestyle;
* Agreeing to follow the constraints generated by the study (presence during the coaching sessions and the final assessment).
* Having signed the informed consent form;
* Social insured;

Exclusion Criteria:

* Presenting a pathology requiring a complementary assessment and/or the implementation of a treatment that could prevent the realization of the coaching or that could modify its effect;
* Subject participating in another clinical study or in period of exclusion from another study;
* Subject deprived of liberty;
* Subject under judicial protection measure;
* Whose main investigator or a qualified co-investigator judges that the state of health or the concomitant treatments are not compatible with the good progress of the clinical study;.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline on quality of life of retired people 12 months after the end of the coaching sessions. | 1 year
  Health quality will be evaluated thanks to a health quality questionnary validated by the World Health Organisation (WHO).

SECONDARY OUTCOMES:
Change from baseline on food behaviors at 1 year after the coaching | 1 year
  Food behaviors will be measure with Balance and dietary diversity questionnaire proposed by the Institut Pasteur de Lille
Change from baseline on food frequency at 1 year after the coaching | 1 year
  Food frequency will be measure with 24-hour reminder of ingestas
  - Visual analogue scales on changes in eating behavior.
Change from baseline on food behavior at 1 year after the coaching | 1 year
  Food behaviors will be measure with Visual analogue scales on changes in eating behavior from 10 (yes really a lot) to 0 (not at all)
Change from baseline on physical activity behaviors at 1 year after the coaching | 1 year
  Visual Analog Scales for Behavioral Change Related to Physical Activity raging from 10 (yes really a lot) to 0 (not at all)
Change from baseline on physical activity frequency at 1 year after the coaching | 1 year
  Marshall Questionnaire for Physical Activity frequency and two questions to evaluate the sedentarity livestyle level.
Change from baseline on endurance at 1 year after the coaching | 1 year
  The using test is :
  • 6 minutes walk test (endurance) Measured in meters
Change from baseline on physical performances (lower limbs) at 1 year after the coaching | 1 year
  The using test is :
  • Stand up chair test to calculate the number of raise on 30 seconds
Change from baseline on physical performances (upper limbs) at 1 year after the coaching | 1 year
  The using test is :
  •Arm curl test to calculate the number of arm bend
Change from baseline on flexibility at 1 year after the coaching | 1 year
  The using test is :
  •Flexible trunk and posterior chain of lower limbs Measured by index ranging from 5 (the palms of the hands touch the ground) to 1 (the fingertips reach the lower shins)
Change from baseline on static balance at 1 year after the coaching | 1 year
  The using test is :
  Unipodal balance (static balance) Measured in seconds
Change from baseline on mobility at 1 year after the coaching | 1 year
  The using test is :
  Get up and go test Measured by index ranging from 5 (the worst) to 1 (the best)
Change from baseline on speed at 1 year after the coaching | 1 year
  The using test is :
  4 meters walking speed
  Measured in seconds
Change from baseline on dynamic balance at 1 year after the coaching | 1 year
  The using test is :
  2 minutes on the spot knee climb This test explores the muscular strength of the lower limbs, dynamic balance and walking Measured in number of knee climb in 2 minutes
Change from baseline on cognitive performances at 1 year after the coaching | 1 year
  Cognitive performances will be measure with :
  - Montreal cognitive assessment test (MOCA test) to evaluate mild cognitive dysfunction
Change from baseline on memory at 1 year after the coaching | 1 year
  It will be measure with :
  - Working Memory Questionnaire
Change from baseline on sleep quality at 1 year after the coaching | 1 year
  It will be measure with :
  - Insomnia Severity Index (ISI) to assess sleep quality
Change from baseline on stress management at 1 year after the coaching | 1 year
  It will be measure with :
  - Cohen's Questionnaire
Change from baseline on anxiety at 1 year after the coaching | 1 year
  It will be measure with :
  - Hospital Anxiety And Depression Queqtionnaire (HAD questionnaire to assess anxiety and depression)
Glucose metabolism | 1 year
  Blood samples will be collected to analyse fasting blood glucose
Lipids metabolism | 1 year
  Blood samples will be collected to analyse: total cholesterol, HDL, LDL, TG
Anthropometric parameters (Body Masse Index) | 1 year
  Weight in kilograms and height in meters will be combined to report BMI in kg/m^2
Anthropometric parameters (waist circumference) | 1 year
  - Waist circumference in centimeters
Body composition | 1 year
  Measurement of body fat by DEXA (Dual X Ray Absorptiometry) for half of the total population :
  * Body fat in grams
  * Lean mass in grams
  * Total mass in grams
  * Visceral fat mass in grams
  * subcutaneous fat mass in grams
  * Bone mineral content in grams
Body composition | 1 year
  Measurement of lean mass by DEXA (Dual X Ray Absorptiometry) for half of the total population :
  * Body fat in percentage
  * Lean mass in percentage
  * Visceral fat mass in percentage
  * subcutaneous fat mass in percentage
Body composition (bone mineral density) | 1 year
  Measurement by DEXA (Dual X Ray Absorptiometry) for half of the total population :
  - Bone mineral density in grams/cm²
Systolic and diastolic blood pressure | 1 year
  Systolic and diastolic blood pressure to calculate blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel LECERF, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: Undecided